# **Section 1: Administrative Information**

Statistical analysis plan (SAP)

Effect of an exercise intervention targeting hip strengthening in patients undergoing revision total hip replacement – A multicenter randomized controlled trial (The Strong Hip Trial)

Martin Bækgaard Stisen<sup>1,2</sup>, Inger Mechlenburg<sup>1,2,3</sup>, and Erik Parner<sup>4</sup>

#### **Affiliations**

# **Trial registration number**

The trial is registered at www.clincaltrials.gov with the number NCT05657054.

#### Version of protocol article used

This SAP was written based on the information in the trial protocol version 1.2, dated 19th of April 2024.

#### **SAP** revision history

No revisions have been made.

# Roles, responsibilities, and signatures

| Role | Name | Date | Signature |
|---|---|---|---|
| Person writing the | Martin Bækgaard Stisen | 15/5/2024 | Martin Stisen |
| SAP | Waitin Bakgaard Stisch | 10/0/2024 | 1 m wi spiser |
| Senior statistician | Erik Parner | 15/5/2024 | Enik Pames |
| responsible | Elik Falliel | | |
| Chief investigator/ | Inger Mechlenburg | 15/5/2024 | Inger Medikeburg |
| Clinical lead | linger Mechienburg | 13/3/2024 | Inger record |
| | | | / 1 |

<sup>&</sup>lt;sup>1</sup>Department of Clinical Medicine, Aarhus University, Aarhus, Denmark.

<sup>&</sup>lt;sup>2</sup>Department of Orthopaedic Surgery, Aarhus University Hospital, Aarhus N, Denmark.

<sup>&</sup>lt;sup>3</sup>Department of Public Health, Section of Sports, Aarhus University, Aarhus, Denmark.

<sup>&</sup>lt;sup>4</sup>Department of Public Health, Section for Biostatistics, Aarhus University, Aarhus, Denmark.

## **Section 2: Introduction**

# **Background and rationale**

Revision total hip replacement (THR) is a common and serious complication after primary THR. In 2022, a total of 1,324 patients underwent revision THR in Denmark (1). Revision THR is commonly undertaken due to loosening, dislocation, fracture, or infection (2,3). Evidence on revision THR in terms of the effectiveness of pain relief and functional improvement is limited (4), and consensus on optimal rehabilitation after revision THR is yet to be established (5). Consequently, there is a need for research exploring different rehabilitation approaches to improve clinical outcomes for patients after revision THR.

Neuromuscular exercise (NEMEX) aims to enhance postural control and functional stability through functional exercises grounded on biomechanical and neuromuscular principles (6). Its effectiveness for reducing pain and improving physical function, and quality of life in hip osteoarthritis (OA) is well-documented (7-10). However, to our knowledge, the effects of postoperatively NEMEX remain unexplored in primary THR patients, as well as in the context of revision THR patients.

Patients with hip OA commonly present with decreased muscle mass and strength (11). These deficiencies persist after primary THR (12-14) and possibly will be even more reduced after revision THR. Notably, muscle strength correlates with functional performance in patients with hip OA (15). Progressive resistance training is considered the most effective intervention for increasing muscle mass and strength (16). Therefore, integrating a resistance training component (external resistance) into the NEMEX program to enhance hip muscle strength and function, seems warranted after revision THR.

#### **Objectives**

The primary objective of this RCT is to compare the effectiveness, four months after initiating rehabilitation, of an exercise intervention targeting hip strengthening (NEMEX-STR) with standard community-based rehabilitation (Usual care) on functional performance in patients undergoing revision THR.

A secondary objective is to compare the effectiveness, 12 months after initiating rehabilitation, on functional performance.

The primary hypothesis for the 4-month and 12-month comparison is that NEMEX-STR is superior to Usual care in functional performance, measured by the 30-second chair stand test (30s-CST).

# **Section 3: Study Methods**

## Trial design

The Strong Hip trial is a multicenter randomized controlled parallel-group assessor-blinded trial conducted across eight hospitals in Denmark, along with their affiliated municipality rehabilitation centers. Participants will be randomized to receive one of two rehabilitation interventions in a 1:1 ratio: either NEMEX-STR or Usual care. The primary outcome is change in functional performance, assessed by the 30s-CST, and the primary endpoint is four months after initiating the rehabilitation intervention. Outcomes will be measured at baseline, as well as at 4- and 12-month follow-ups. Detailed descriptions of the rehabilitation exercise protocols can be found in the trial protocol.

Reporting of the trial will follow the 'Consolidated Standards of Reporting Trials' (CONSORT) statement guidelines (17). This SAP is reported following the 'Guidelines for the Content of Statistical Analysis Plan in Clinical Trials' (18).

#### **Randomization**

Following their revision THR, patients are randomized in a 1:1 ratio to either NEMEX-STR or Usual care. Utilizing the Research Electronic Data Capture (REDCap) randomize tool, a computer-generated list of random numbers is generated (19). Randomization is stratified by the participating hospitals with block sizes selected randomly. Throughout the trial, block sizes and randomization sequences remain blinded for the administrator of the randomization procedure.

#### Sample size

The sample size calculation is based on the expected between-group difference in the 30s-CST from baseline to 4-month follow-up. Given the absence of revision THR-specific data, the calculation relies on primary hip and knee replacement studies, as well as data from patients with hip and knee OA. The major clinically important improvement for 30s-CST among hip OA patients is defined as 2.1 chair stands (20). Mikkelsen et al. (21) observed a mean change of 2.84 chair stands in patients undergoing primary THR following 10 weeks of supervised progressive resistance training in combination with unsupervised home-based exercise. Further, Abbott et al. (22) reported a mean change of 0.59 among patients with hip or knee OA at 1-year follow-up after receiving usual care. The standard deviation for the 30s-CST, obtained from the 95% CI of the change in the intervention group of the study by Mikkelsen et al. (21), is calculated as 3.03. With a significance level set at 5% and a sample size of 60 patients, the study will have 80% power to detect a change of 2.25 chair stands. Accounting

for loss to follow-up of 40%, determined in consideration of the complex population, the total sample

size is 84 patients.

**Framework** 

The overall objective of this trial is to ascertain whether NEMEX-STR results in a clinically and

statistically significantly greater improvement compared to Usual care in the 30s-CST, Hip Disability

and Osteoarthritis Outcome Score (HOOS), 40m Fast-paced Walk Test (40m-FPWT), 9-step Timed

Stair Climb Test (9-step TSCT), Leg Extensor Power, Global perceived effect (GPE), Adverse events

and serious adverse events, Adherence and drop-outs, The International Physical Activity Question-

naire (IPAQ), Numerical rating scale for pain (NRS), and European Quality of Life - 5 Dimensions

(EQ-5D-5L). The primary hypothesis is that NEMEX-STR is superior to Usual care at 4 months, and

the secondary hypothesis is that NEMEX-STR is superior to Usual care at 12 months.

Statistical interim analysis and stopping guidance

No formal statistical interim analysis is planned for the StrongHip Trial. Participant enrolment started

in November 2022 and is expected to be completed by June 2024. All participants are expected to

have completed 4-month follow-up assessments by February 2025, and 12-month follow-up assess-

ments by October 2025.

Timing of final analysis

For the 4-month comparison, the final analysis is planned to be conducted when all randomized par-

ticipants have completed the 4-month follow-up. The anticipated publication submission time is ul-

timo 2025. Likewise, for the 12-month comparison, the final analysis is planned when all randomized

participants have completed the 12-month follow-up. The anticipated publication submission time is

ultimo 2026.

Timing of outcome assessments

This trial entails outcome assessments at three time points; baseline, 4 months after initiation of the

rehabilitation intervention, and 12 months after initiation of the rehabilitation intervention. An over-

view of the timing of outcome assessments is presented in Table 1.

|4

# **Section 4: Statistical Principles**

#### Confidence intervals and P values

All statistical tests and confidence intervals will be two-sided. The statistical level of significance will be set to 0.05 and outcomes will be presented with 95% confidence intervals.

#### Adherence and protocol deviations

For the NEMEX-STR group, adherence to exercise will be self-registered by the participants in an exercise log (supervised sessions will be registered by the physiotherapists supervising the exercise sessions). Adherence will be presented as descriptive statistics (numbers and percentages). Adherence percentage is calculated as the number of sessions completed divided by the number of sessions planned multiplied by 100%. High adherence for the 4 months is defined as attendance in  $\geq$ 80% of the exercise sessions. Further, for the NEMEX-STR group, the proportion of patients reaching difficulty levels 1, 2, and 3 will be presented. Any protocol deviations, i.e., drop-outs, reoperation, or initiation of other exercise treatments, will also be presented as descriptive statistics (numbers and percentages).

# **Analysis populations**

The primary analyses will follow the Intention-to-Treat (ITT) principle, encompassing all participants randomized to treatment in the analyses, irrespective of adherence or protocol deviations. Participants who drop out will contribute data to their respective allocation groups until they drop out, without any imputations made.

A secondary analysis will incorporate a per-protocol analysis, wherein per protocol is defined as patients complying with the assigned treatment.

Subsequent per-protocol analyses will be conducted, excluding patients with poor adherence to the exercise sessions in the NEMEX-STR intervention (<80% of the planned sessions), and participants in the Usual care intervention who deviate from the randomized treatment.

# **Section 5: Trial Population**

#### Screening data

At each of the eight hospitals, eligible revision THR patients will be screened for the predetermined eligibility criteria. Patients meeting these criteria will be invited to participate. The count of patients

who does not meet the criteria and the reason for ineligibility will be documented in a CONSORT flow chart (Figure 1).

# **Eligibility**

Participants meeting the following inclusion and exclusion criteria are considered eligible for this trial.

#### Inclusion criteria:

- 1. Undergoing first revision THR.
- 2. Age  $\geq$ 18 years.
- 3. Acceptance to participate in an exercise program for 16 weeks.
- 4. Cup and/or stem replaced, or a combination of liner and caput replaced.
- 5. Able to perform baseline tests.

#### Exclusion criteria:

- 1. Dependency on a wheelchair.
- 2. Other preplanned lower limb surgery within 12 months.
- 3. Body Mass Index (BMI) score >40.
- 4. Currently undergoing cancer treatment, e.g., chemo-, immuno-, or radiotherapy.
- 5. Comorbidities that prevent exercise, e.g. stroke, significant heart diseases, or similar (Orthopedic surgeons and/or physiotherapists determine if a patient is unable to exercise during consultations or upon discovering comorbidities).
- 6. Inadequacy in written and spoken Danish.
- 7. Mentally unable to participate.

# Recruitment

The CONSORT flowchart will present the total number of patients who were screened, excluded (with reasons), randomized, receiving allocated treatment, discontinued intervention (with reasons), lost to follow-up (with reasons), included in the ITT analysis, and included in the per-protocol analysis.

#### Withdrawal/follow-up

Participants are allowed to withdraw from the study at any time during the trial period. Withdrawn participants will be encouraged to complete outcome assessments even though they stop attending exercise sessions. Withdrawals will be categorized into two options; [1] complete withdrawal from

the trial without further outcome assessments, and [2] withdrawal from the exercise intervention

while still attending outcomes assessments. The reason and timing of withdrawals and loss to follow-

up will be outlined in the CONSORT flowchart.

**Baseline participant characteristics** 

Baseline participant characteristics will be presented by randomization group as seen in Table 2,

entailing the following information: Gender, age, height, weight, cohabiting status, educational level,

employment status, number of comorbidities measured with the Charlson Comorbidity Index, anal-

gesic use (type(s) and frequency), indication for revision THR, time since primary THR, indication

for primary THR, and indication for revision THR. Continuous variables will be presented as either

mean with standard deviation (SD) if normally distributed, or as median with interquartile range

(IQR) if not normally distributed. For categorical variables, numbers and corresponding percentages

will be presented.

**Section 6: Analysis** 

**Outcome definitions** 

Primary outcome

30s Chair Stand Test (30s-CST)

The primary outcome is between-group differences in change from baseline to 4 months in the 30s-

CST, measured by the number of repetitions (20,23,24). The 30s-CST was selected as the primary

outcome because it is an objective measure of lower-extremity muscle strength and functional per-

formance, which is simply standardized between testers and test locations, and considered valid and

reliable (20,25,26). The 30s-CST is recommended by the Osteoarthritis Research Society Interna-

tional (OARSI) as part of the minimum core set of performance-based tests of physical function in

people diagnosed with hip OA or following joint replacement (27).

Given the absence of a minimal important change (MIC) established specifically for the 30s-CST

for revision THR patients, we will calculate a trial-specific MIC by subtracting the mean score of

participants who reported experiencing a 'small but not important improvement' in the Global Per-

ceived Effect (GPE) from the mean score of those reporting an 'important improvement' in the GPE.

| 7

# Secondary outcomes

Hip Disability and Osteoarthritis Outcome Score (HOOS)

As a secondary outcome measure, the study will examine the between-group differences in change from baseline to 4 and 12 months in the five separate subscales of the HOOS covering pain, symptoms, activity limitations daily living, sport and recreation function, and hip-related quality of life HOOS (28). Each subscale ranges from 0-100, worst to best (29). It is valid and reliable in patients undergoing THR (28,30,31).

The 40m Fast-paced Walk Test (40m-FPWT)

Another secondary outcome of interest is the between-group differences in change from baseline to 4 and 12 months in the 40m-FPWT, quantified in seconds. It is measured as the time it takes to walk a 10m walkway four times in total as quickly and as safely as possible (20,23). The 40m-FPWT is a valid measure of maximum walking speed over a short distance, exhibiting excellent reliability (20).

The 9-step Timed Stair Climb Test (9-step TSCT)

Another secondary outcome is the between-group differences in change from baseline to 4 and 12 months in the 9-step TSCT, measured in seconds (23,32). It is measured as the time it takes to ascend and descend a 9-step stair and has excellent reliability in patients with hip OA (20,33-35).

Nottingham Leg Extensor Power Rig (NLEPR)

Another secondary outcome is the between-group differences in change from baseline to 4 and 12 months in leg extensor muscle power (watt/kg), measured with the NLEPR. Leg extensor muscle power is highly correlated with functional performance (36-38), and the NLEPR has acceptable reliability in patients undergoing THR (33,39,40).

Global perceived effect (GPE)

Another secondary outcome is the proportion of participants in each treatment group experiencing an 'important improvement' at 4 and 12 months using the GPE. It will be assessed for three domains; pain, activities of daily living, and quality of life rated on a 7-point Likert scale (41,42).

Adverse events and serious adverse events

Adverse events (AE) and serious adverse events (SAE) will be continuously recorded throughout the trial and defined in accordance with the 'International Council on Harmonisation of Technical Re-

quirements for Pharmaceuticals for Human Use - Guideline for good clinical practice' (43,44). Physiotherapists supervising the exercise sessions will monitor the events, and patients will be asked about potential AE and SAE during follow-ups following recommendations from the CONSORT group.

Adherence and drop-outs

Exercise adherence and progression within the NEMEX-STR intervention will be documented by the supervising physiotherapist. Further, patients will maintain exercise logs, to monitor adherence to home-based sessions. Adherence is described in detail in the 'Adherence and protocol deviations' section.

#### Other outcomes

Physical activity

An other outcome of interest is physical activity assessed by the International Physical Activity Questionnaire (IPAQ), which is a 7-item questionnaire containing open-ended questions about the patient's last 7-day recall of physical activity (45,46).

Numerical rating scale for pain (NRS)

An other outcome is patient-reported pain intensity at rest rated using NRS, which is an 11-item scale ranging from 0 to 10, with 0 indicating no pain and 10 indicating the worst imaginable pain (47,48).

European Quality of Life - 5 Dimensions (EQ-5D-5L)

An other outcome is Health-Related Quality of Life evaluated through the EQ-5D-5L, a patient-reported instrument that encompasses five dimensions; mobility, self-care, usual daily activities, pain/discomfort, and anxiety/depression (49). Additionally, it includes a visual analog scale (VAS) to measure self-rated health. The EQ-5D-5L is a valid and reliable measure of HRQoL in patients undergoing primary THR (49-51).

# **Analysis methods**

Between-group comparisons of changes from baseline to follow-up in both the primary and continuous secondary outcomes will be analyzed following the ITT principle (i.e., patients analyzed according to their initial randomization, irrespective of adherence or potential crossovers) using a mixed-effects model of baseline and follow-up measurements as outcome, but restricting the mean baseline measurement to be the same in the two randomization groups (52,53). Fixed effects will

Date: 15.05.2024

Version 1.0

encompass the treatment group and time point, allowing evaluation of the effects of both interven-

tions and observing progression over time. To accommodate within-patient correlation and poten-

tial clustering effects, random effects for patients and hospital sites will be incorporated. Further,

fixed covariates such as age and sex, will be included to minimize the residual variation.

Missing data

As stated prior, no imputations will be applied in the analysis. However, the mixed-effects model

manages potential missing outcome data. Each randomized participant will be included in the ITT

analysis with the data collected for that participant. An effort to collect data from all randomized

participants will be made, regardless of their adherence to interventions.

Additional analysis

No additional analyses are planned for the 4- and 12-month follow-up.

Harms

Adverse events and serious adverse events will be presented as numbers and percentages for each

event.

**Statistical software** 

All statistical analyses will be conducted using Stata (StataCorp, College Station, Texas, USA).

| 10

#### References

- 1. Danish Hip Arthroplasty Register. Annual Reports 2022. 2022.
- 2. Karachalios T, Komnos G, Koutalos A. Total hip arthroplasty: Survival and modes of failure. EFORT open reviews 2018; 3: 232-239.
- 3. Ulrich SD, Seyler TM, Bennett D, Delanois RE, Saleh KJ, Thongtrangan I, et al. Total hip arthroplasties: what are the reasons for revision? International orthopaedics 2008; 32: 597-604.
- 4. Singh JA, Lewallen DG. Patient-level clinically meaningful improvements in activities of daily living and pain after total hip arthroplasty: data from a large US institutional registry. Rheumatology (Oxford, England) 2013; 52: 1109-1118.
- 5. Newman M, Barker K. Rehabilitation of revision total hip replacement: A multi-centre survey of current practice. Musculoskeletal care 2017; 15: 386-394.
- 6. Ageberg E, Roos EM. Neuromuscular exercise as treatment of degenerative knee disease. Exerc Sport Sci Rev 2015; 43: 14-22.
- 7. Ageberg E, Link A, Roos EM. Feasibility of neuromuscular training in patients with severe hip or knee OA: The individualized goal-based NEMEX-TJR training program. BMC musculoskeletal disorders 2010; 11: 126.
- 8. Ageberg E, Nilsdotter A, Kosek E, Roos EM. Effects of neuromuscular training (NEMEX-TJR) on patient-reported outcomes and physical function in severe primary hip or knee osteoarthritis: a controlled before-and-after study. BMC musculoskeletal disorders 2013; 14: 232.
- 9. Villadsen A, Overgaard S, Holsgaard-Larsen A, Christensen R, Roos EM. Postoperative effects of neuromuscular exercise prior to hip or knee arthroplasty: a randomised controlled trial. Annals of the rheumatic diseases 2014; 73: 1130-1137.
- 10. Villadsen A, Overgaard S, Holsgaard-Larsen A, Christensen R, Roos EM. Immediate efficacy of neuromuscular exercise in patients with severe osteoarthritis of the hip or knee: a secondary analysis from a randomized controlled trial. The Journal of rheumatology 2014; 41: 1385-1394.
- 11. Loureiro A, Mills PM, Barrett RS. Muscle weakness in hip osteoarthritis: a systematic review. Arthritis care & research 2013; 65: 340-352.
- 12. Winther SB, Husby VS, Foss OA, Wik TS, Svenningsen S, Engdal M, et al. Muscular strength after total hip arthroplasty. A prospective comparison of 3 surgical approaches. Acta orthopaedica 2016; 87: 22-28.
- 13. Rasch A, Byström AH, Dalén N, Martinez-Carranza N, Berg HE. Persisting muscle atrophy two years after replacement of the hip. The Journal of bone and joint surgery British volume 2009; 91: 583-588.
- 14. Rasch A, Dalén N, Berg HE. Muscle strength, gait, and balance in 20 patients with hip osteoarthritis followed for 2 years after THA. Acta orthopaedica 2010; 81: 183-188.
- 15. Bieler T, Magnusson SP, Christensen HE, Kjaer M, Beyer N. Muscle power is an important measure to detect deficits in muscle function in hip osteoarthritis: a cross-sectional study. Disability and rehabilitation 2017; 39: 1414-1421.

16. American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc 2009; 41: 687-708.

- 17. Moher D, Hopewell S, Schulz KF, Montori V, Gøtzsche PC, Devereaux PJ, et al. CONSORT 2010 Explanation and Elaboration: updated guidelines for reporting parallel group randomised trials. 2010; 340: c869.
- 18. Gamble C, Krishan A, Stocken D, Lewis S, Juszczak E, Doré C, et al. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. Jama 2017; 318: 2337-2343.
- Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)—A metadata-driven methodology and workflow process for providing translational research informatics support. Journal of Biomedical Informatics 2009; 42: 377-381.
- 20. Wright AA, Cook CE, Baxter GD, Dockerty JD, Abbott JH. A comparison of 3 methodological approaches to defining major clinically important improvement of 4 performance measures in patients with hip osteoarthritis. J Orthop Sports Phys Ther 2011; 41: 319-327.
- 21. Mikkelsen LR, Mechlenburg I, Søballe K, Jørgensen LB, Mikkelsen S, Bandholm T, et al. Effect of early supervised progressive resistance training compared to unsupervised homebased exercise after fast-track total hip replacement applied to patients with preoperative functional limitations. A single-blinded randomised controlled trial. Osteoarthritis and cartilage 2014; 22: 2051-2058.
- 22. Abbott JH, Robertson MC, Chapple C, Pinto D, Wright AA, Leon de la Barra S, et al. Manual therapy, exercise therapy, or both, in addition to usual care, for osteoarthritis of the hip or knee: a randomized controlled trial. 1: clinical effectiveness. Osteoarthritis and cartilage 2013; 21: 525-534.
- 23. Bennell K, Dobson F, Hinman R. Measures of physical performance assessments: Self-Paced Walk Test (SPWT), Stair Climb Test (SCT), Six-Minute Walk Test (6MWT), Chair Stand Test (CST), Timed Up & Go (TUG), Sock Test, Lift and Carry Test (LCT), and Car Task. Arthritis care & research 2011; 63 Suppl 11: S350-370.
- 24. Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport 1999; 70: 113-119.
- 25. Gill SD, de Morton NA, Mc Burney H. An investigation of the validity of six measures of physical function in people awaiting joint replacement surgery of the hip or knee. Clinical rehabilitation 2012; 26: 945-951.
- 26. Gill S, McBurney H. Reliability of performance-based measures in people awaiting joint replacement surgery of the hip or knee. Physiother Res Int 2008; 13: 141-152.
- 27. Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, et al. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis and cartilage 2013; 21: 1042-1052.
- 28. Nilsdotter AK, Lohmander LS, Klässbo M, Roos EM. Hip disability and osteoarthritis outcome score (HOOS)--validity and responsiveness in total hip replacement. BMC musculoskeletal disorders 2003; 4: 10.

29. Nilsdotter A, Bremander A. Measures of hip function and symptoms: Harris Hip Score (HHS), Hip Disability and Osteoarthritis Outcome Score (HOOS), Oxford Hip Score (OHS), Lequesne Index of Severity for Osteoarthritis of the Hip (LISOH), and American Academy of Orthopedic Surgeons (AAOS) Hip and Knee Questionnaire. Arthritis care & research 2011; 63 Suppl 11: S200-207.

- 30. Thorborg K, Roos EM, Bartels EM, Petersen J, Hölmich P. Validity, reliability and responsiveness of patient-reported outcome questionnaires when assessing hip and groin disability: a systematic review. Br J Sports Med 2010; 44: 1186-1196.
- 31. Klässbo M, Larsson E, Mannevik E. Hip disability and osteoarthritis outcome score. An extension of the Western Ontario and McMaster Universities Osteoarthritis Index. Scand J Rheumatol 2003; 32: 46-51.
- 32. Perron M, Malouin F, Moffet H. Assessing advanced locomotor recovery after total hip arthroplasty with the timed stair test. Clinical rehabilitation 2003; 17: 780-786.
- 33. Bieler T, Magnusson SP, Kjaer M, Beyer N. Intra-rater reliability and agreement of muscle strength, power and functional performance measures in patients with hip osteoarthritis. Journal of rehabilitation medicine 2014; 46: 997-1005.
- 34. Kennedy DM, Stratford PW, Wessel J, Gollish JD, Penney D. Assessing stability and change of four performance measures: a longitudinal study evaluating outcome following total hip and knee arthroplasty. BMC musculoskeletal disorders 2005; 6: 3-3.
- 35. C. Davey R, Edwards SM, Cochrane T. Test–retest Reliability of Lower Extremity Functional and Self-reported Measures in Elderly with Osteoarthritis. Advances in Physiotherapy 2003; 5: 155-160.
- 36. Foldager F, Jørgensen PB, Tønning LU, Petersen ET, Jakobsen SS, Vainorius D, et al. The relationship between muscle power, functional performance, accelerometer-based measurement of physical activity and patient-reported outcomes in patients with hip osteoarthritis: A cross-sectional study. Musculoskeletal Science and Practice 2022; 62: 102678.
- 37. Bean JF, Leveille SG, Kiely DK, Bandinelli S, Guralnik JM, Ferrucci L. A comparison of leg power and leg strength within the InCHIANTI study: which influences mobility more? J Gerontol A Biol Sci Med Sci 2003; 58: 728-733.
- 38. Foldvari M, Clark M, Laviolette LC, Bernstein MA, Kaliton D, Castaneda C, et al. Association of muscle power with functional status in community-dwelling elderly women. J Gerontol A Biol Sci Med Sci 2000; 55: M192-199.
- 39. Mikkelsen LR, Mikkelsen S, Søballe K, Mechlenburg I, Petersen AK. A study of the inter-rater reliability of a test battery for use in patients after total hip replacement. Clinical rehabilitation 2015; 29: 165-174.
- 40. Bassey EJ, Short AH. A new method for measuring power output in a single leg extension: feasibility, reliability and validity. Eur J Appl Physiol Occup Physiol 1990; 60: 385-390.
- 41. Kamper SJ, Ostelo RW, Knol DL, Maher CG, de Vet HC, Hancock MJ. Global Perceived Effect scales provided reliable assessments of health transition in people with musculoskeletal disorders, but ratings are strongly influenced by current status. Journal of clinical epidemiology 2010; 63: 760-766.e761.

42. Fitzgerald GK, Hinman RS, Zeni J, Jr., Risberg MA, Snyder-Mackler L, Bennell KL. OARSI Clinical Trials Recommendations: Design and conduct of clinical trials of rehabilitation interventions for osteoarthritis. Osteoarthritis and cartilage 2015; 23: 803-814.

- 43. Schulz KF, Altman DG, Moher D. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. Trials 2010; 11: 32.
- 44. Ioannidis JP, Evans SJ, Gøtzsche PC, O'Neill RT, Altman DG, Schulz K, et al. Better reporting of harms in randomized trials: an extension of the CONSORT statement. Ann Intern Med 2004; 141: 781-788.
- 45. Craig CL, Marshall AL, Sjöström M, Bauman AE, Booth ML, Ainsworth BE, et al. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc 2003; 35: 1381-1395.
- 46. Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the international physical activity questionnaire short form (IPAQ-SF): A systematic review. International Journal of Behavioral Nutrition and Physical Activity 2011; 8: 115.
- 47. Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis care & research 2011; 63: S240-S252.
- 48. Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, et al. Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage 2011; 41: 1073-1093.
- 49. Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, et al. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res 2011; 20: 1727-1736.
- 50. Conner-Spady BL, Marshall DA, Bohm E, Dunbar MJ, Noseworthy TW. Comparing the validity and responsiveness of the EQ-5D-5L to the Oxford hip and knee scores and SF-12 in osteoarthritis patients 1 year following total joint replacement. Qual Life Res 2018; 27: 1311-1322.
- 51. Conner-Spady BL, Marshall DA, Bohm E, Dunbar MJ, Loucks L, Al Khudairy A, et al. Reliability and validity of the EQ-5D-5L compared to the EQ-5D-3L in patients with osteoarthritis referred for hip and knee replacement. Qual Life Res 2015; 24: 1775-1784.
- 52. Liu GF, Lu K, Mogg R, Mallick M, Mehrotra DV. Should baseline be a covariate or dependent variable in analyses of change from baseline in clinical trials? Stat Med 2009; 28: 2509-2530.
- 53. Liang K-Y, Zeger SL. Longitudinal Data Analysis of Continuous and Discrete Responses for Pre-Post Designs. Sankhyā: The Indian Journal of Statistics, Series B (1960-2002) 2000; 62: 134-148.

# Figures and tables



**FIGURE 1.** Flow chart with expected enrolment, randomization, and follow-up. Abbreviations: THR, Total Hip Replacement; 30s-CST, 30-second Chair Stand Test.



**FIGURE 2.** Change in 30-second chair stand test from baseline to 4-month follow-up. This figure is an example and displays the anticipated changes. Abbreviations: 30s-CST, 30s Chair Stand Test.



**FIGURE 3.** The proportion of participants reaching the clinically relevant improvement in primary and secondary outcomes. This figure is an example and displays the anticipated changes.

Abbreviations: MIC, Minimal Important Change; 30s-CST, 30s Chair Stand Test; 40m-FPWT, 40m Fast-paced Walk Test; 9-step TSCT, 9-step Timed Stair Climb Test; HOOS, Hip Disability and Osteoarthritis Outcome Score; ADL, Activity Limitations Daily Living; QoL, Quality of Life.



**FIGURE 4.** Change in 30-second chair stand test from baseline to 4- and 12-month follow-up. This figure is an example and displays the anticipated changes. Abbreviations: 30s-CST, 30s Chair Stand Test.

**TABLE 1.** Table of outcome and baseline characteristics assessments

| Assessments | Baseline | 4 months | 12 months |
|-------------------------------------------|----------|----------|-----------|
| Primary outcome | | | |
| 30s Chair Stand Test | X | X | X |
| Secondary outcomes | | | |
| HOOS | X | X | X |
| 40m Fast-paced Walk Test | X | X | X |
| 9-step Timed Stair Climb Test | X | X | X |
| Leg extension muscle power | X | X | X |
| Global perceived effect | | Χ | Χ |
| Adverse events and serious adverse events | | X | X |
| Adherence and drop-outs | | X | |
| Other outcomes | | | |
| IPAQ | Χ | X | X |
| Pain (NRS) | Χ | X | X |
| EQ-5D-5L | Χ | X | X |
| Baseline characteristics | | | |
| Gender | Χ | | |
| Age | Χ | | |
| Height | X | | |
| Weight | X | | |
| Cohabiting status | X | | |
| Highest obtained educational level | Χ | | |
| Employment status | X | | |
| Number of comorbidities | X | | |
| Analgesic use | X | | |
| Indication for revision THR | X | | |
| Time since primary THR | X | | |
| Indication for primary THR | Χ | | |

Abbreviations: HOOS, Hip Disability and Osteoarthritis Outcome Score; IPAQ, The International Physical Activity Questionnaires; NRS, Numeric Rating Scale; EQ-5D-5L, European Quality of Life - 5 Dimensions; THR, Total Hip Replacement.

**TABLE 2.** Baseline characteristics.

Characteristic NEMEX-STR (n=) Usual care (n=) Gender, n(%) Female Male Mean age (SD), y Mean BMI (SD), kg/m<sup>2</sup> Cohabiting status, n(%) Cohabiting Living alone Educational level, n(%) Primary school High school or similar Vocational education Higher education Employment status, n(%) Employed or self-employed Unemployed Retired Comorbidities (CCI), n(%) Low Medium High Analgesic use, n(%) Acetaminophen Nonsteroidal anti-inflammatory drugs Morphine or opioids Other Analgesic use frequency, n(%) Never Monthly Weekly Daily Indication for revision THR, n(%) Implant wear Loosening Dislocation or hip instability Pain Infection Fracture Other Time since primary THR (SD), y Indication for primary THR, n(%) Osteoarthritis Fracture Dislocation Other types of arthritis Congenital hip problems Other

Abbreviations: BMI, Body Mass Index; CCI, Charlson Comorbidity Index; THR, Total Hip Replacement

**TABLE 3.** Change from baseline to 4-month follow-up in primary and secondary outcomes.

| The state of the s | | NEMEX-STR | | | Usual care | | Difference in change |
|---|---|---|---|---|---|---|---|
| Intention to treat analysis | | | | | | | |
| | Baseline<br>(SD) | 4-month<br>(SD) | Change<br>(CI) | Baseline<br>(SD) | 4-month<br>(SD) | Change<br>(CI) | Difference<br>(CI) |
| Functional performance 30s-CST 40m-FPWT 9-step TSCT Leg Extension Power Patient-reported outcomes HOOS Symptoms HOOS Pain HOOS ADL HOOS Sport/recreation HOOS Hip-related QoL | | | | | | | |
| | | Per-p | rotocol analy | sis | | | |
| | Baseline<br>(SD) | 4-month<br>(SD) | Change<br>(CI) | Baseline<br>(SD) | 4-month<br>(SD) | Change<br>(CI) | Difference<br>(CI) |
| Functional performance 30s-CST 40m-FPWT 9-step TSCT Leg Extension Power Patient-reported outcomes HOOS Symptoms HOOS Pain HOOS ADL HOOS Sport/recreation HOOS Hip-related QoL | | | | | | | |

Abbreviations: 30s-CST, 30s Chair Stand Test; 40m-FPWT, 40m Fast-paced Walk Test; 9-step TSCT, 9-step Timed Stair Climb Test; HOOS, Hip Disability and Osteoarthritis Outcome Score; ADL, Activity Limitations Daily Living; QoL, Quality of Life.

**TABLE 4**. Serious adverse events, adverse events, drop-outs, and adherence to interventions at 4-month follow-up.

| | NEMEX-STR | Usual care |
|---------------------------------------|-------------------|-------------|
| Serious adverse events – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Adverse events – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Drop-outs – n (%) | | |
| Mean adherence to exercise – (%)* | | |
| ≥ 80% adherence – n (%) | | |
| ≥ 50% adherence – n (̇%́) | | |
| < 50% adherence – n (%) | | |
| Adherence to Usual care** - n (%) | | |
| *Adherence to evercise: Number of nat | ients in the NEME | X-STR group |

<sup>\*</sup>Adherence to exercise; Number of patients in the NEMEX-STR group who participated in  $\geq$  80%,  $\geq$  50%, < 50% of exercise sessions.

<sup>\*\*</sup>Adherence to Usual care; Number of patients in the Usual care group who followed the exercise regimen and didn't crossover to other exercise treatments.

**TABLE 5.** Change from baseline to 12-month follow-up in primary and secondary outcomes.

| | | NEMEX-STR | | | Usual care | | Difference in change |
|---|---|---|---|---|---|---|---|
| Intention to treat analysis | | | | | | | |
| | Baseline<br>(SD) | 12-month<br>(SD) | Change<br>(CI) | Baseline<br>(SD) | 12-month<br>(SD) | Change<br>(CI) | Difference<br>(CI) |
| Functional performance 30s-CST 40m-FPWT 9-step TSCT Leg Extension Power Patient-reported outcomes HOOS Symptoms HOOS Pain HOOS ADL HOOS Sport/recreation HOOS Hip-related QoL | | | | | | | |
| | | Per-p | rotocol analy | sis | | | |
| | Baseline<br>(SD) | 12-month<br>(SD) | Change<br>(CI) | Baseline<br>(SD) | 12-month<br>(SD) | Change<br>(CI) | Difference<br>(CI) |
| Functional performance 30s-CST 40m-FPWT 9-step TSCT Leg Extension Power Patient-reported outcomes HOOS Symptoms HOOS Pain HOOS ADL HOOS Sport/recreation HOOS Hip-related QoL | | | | | | | |

Abbreviations: 30s-CST, 30s Chair Stand Test; 40m-FPWT, 40m Fast-paced Walk Test; 9-step TSCT, 9-step Timed Stair Climb Test; HOOS, Hip Disability and Osteoarthritis Outcome Score; ADL, Activity Limitations Daily Living; QoL, Quality of Life.

**TABLE 6**. Serious adverse events, adverse events, and drop-outs at 12-month follow-up.

| · | NEMEX-STR | Usual care |
|--------------------------------|-----------|------------|
| Serious adverse events – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Adverse events – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Specification – n (%) | | |
| Drop-outs – n (%) | | |